CLINICAL TRIAL: NCT03009643
Title: Salvage Treatment of Inhaled Nitric Oxide in Patients With Refractory Hypoxemia After Aortic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Guowei Tu, Attending doctor, Department of cardiac surgery intensive care unit, Principal Investigator, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STiNO
Record Dates: First submitted 2016-12-26; First posted 2017-01-04 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Nitric Oxide; Hypoxemia; Aortic Surgery
Keywords: Nitric Oxide; hypoxemia; aortic surgery
MeSH Terms: conditions — Hypoxia | interventions — Hemodynamic Monitoring

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- iNO Group (Experimental): Patients are treated with iNO at a concentration of 5-10 ppm for 3-5 days according to the clinical conditions
  Interventions: Drug: Inhaled Nitric Oxide; Device: lung protective mechanical ventilation; Device: Hemodynamic monitoring
- Control (Other): Patients are treated without iNO.
  Interventions: Device: lung protective mechanical ventilation; Device: Hemodynamic monitoring

INTERVENTIONS:
Drug: Inhaled Nitric Oxide — Patients are treated with iNO for 3-5 days.The concentration of inhaled Nitric Oxide is around 5-10ppm.
  Arms: iNO Group
Device: lung protective mechanical ventilation — Mechanical ventilation in the SIMV mode (ventilators Evita 2 or 4,Dräger, Lübeck, Germany) with VT 6-8ml/kg
Device: Hemodynamic monitoring — Flotrac/Vigileo (Edwards Lifesciences) are used to guide the fluid management.

SUMMARY:
Hypoxemia is a common complication after aortic surgery. As this complication has an adverse effect on the postoperative course of the patient, early treatment is important; however, the mechanism of hypoxemia after surgery for acute aortic dissection remains unclear. Recently, the investigators found that inhaled Nitric Oxide can improve the oxygenation in some of these patients. The investigators are trying to evaluate the effectiveness and safety of inhaled Nitric Oxide in patients with refractory hypoxemia after aortic surgery.

DETAILED DESCRIPTION:
Several risk factors for severe hypoxemia after aortic surgery have been reported including advanced age, obesity, smoking history, previous heart surgery,emergency surgery,reduced cardiac function, advanced chronic obstructive pulmonary disease, excessive volume of blood transfusion,and prolonged CPB time. The routine treatment includes lung protective mechanical ventilation, recruitment maneuvers and glucocorticoids.

No previous clinical studies have reported the effectiveness and safety of inhaled Nitric Oxide in patients with refractory hypoxemia after aortic surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with refractory hypoxemia after aortic surgery;
2. Accepting invasive mechanical ventilation;
3. Chest X-ray and lung ultrasound to exclude the respiratory factors (eg. pulmonary edema, obstructive atelectasis, pleural effusion, pneumothorax) and hemodynamic factors (pericardial tamponade, acute pulmonary hypertension, intracardiac shunt);
4. The ventilator parameters: PEEP>10cmH2O, VT 6-8ml/kg;
5. The PaO2/FiO2 <= 100mmHg.

Exclusion Criteria:

1. Age <18 years old;
2. Pregnant women;
3. Past medical history included COPD or mental illness;
4. The serious infection or sepsis patients;
5. Patients with pulmonary hypertension and right ventricular dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-10; Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Mechanical ventilation time (days) | During whole ICU stay. From date of randomization until the date of death or discharge from ICU, up to 6 months.

SECONDARY OUTCOMES:
ICU mortality | From date of randomization until the date of death or discharge from ICU, up to 6 months.
length of hospital stay (days) | From date of randomization until the date of death or discharge from hospital, up to 6 months.
length of ICU stay (days) | From date of randomization until the date of death or discharge from ICU, up to 6 months.
hospital mortality | From date of randomization until the date of death or discharge from hospital, up to 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Zhe Luo, PhD, Study Director — Department of Critical Care Medicine
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garcia-Delgado M, Navarrete-Sanchez I, Colmenero M. Preventing and managing perioperative pulmonary complications following cardiac surgery. Curr Opin Anaesthesiol. 2014 Apr;27(2):146-52. doi: 10.1097/ACO.0000000000000059. PMID 24514031
- [Background] Ball L, Battaglini D, Pelosi P. Postoperative respiratory disorders. Curr Opin Crit Care. 2016 Aug;22(4):379-85. doi: 10.1097/MCC.0000000000000312. PMID 27168252
- [Background] Griffiths MJ, Evans TW. Inhaled nitric oxide therapy in adults. N Engl J Med. 2005 Dec 22;353(25):2683-95. doi: 10.1056/NEJMra051884. No abstract available. PMID 16371634
- [Result] Nakajima T, Kawazoe K, Izumoto H, Kataoka T, Niinuma H, Shirahashi N. Risk factors for hypoxemia after surgery for acute type A aortic dissection. Surg Today. 2006;36(8):680-5. doi: 10.1007/s00595-006-3226-5. PMID 16865510
- [Result] Wang Y, Xue S, Zhu H. Risk factors for postoperative hypoxemia in patients undergoing Stanford A aortic dissection surgery. J Cardiothorac Surg. 2013 Apr 30;8:118. doi: 10.1186/1749-8090-8-118. PMID 23631417
- [Result] Palmer RM, Ferrige AG, Moncada S. Nitric oxide release accounts for the biological activity of endothelium-derived relaxing factor. Nature. 1987 Jun 11-17;327(6122):524-6. doi: 10.1038/327524a0. PMID 3495737
- [Result] Frostell C, Fratacci MD, Wain JC, Jones R, Zapol WM. Inhaled nitric oxide. A selective pulmonary vasodilator reversing hypoxic pulmonary vasoconstriction. Circulation. 1991 Jun;83(6):2038-47. doi: 10.1161/01.cir.83.6.2038. PMID 2040056
- [Result] Frostell CG, Blomqvist H, Hedenstierna G, Lundberg J, Zapol WM. Inhaled nitric oxide selectively reverses human hypoxic pulmonary vasoconstriction without causing systemic vasodilation. Anesthesiology. 1993 Mar;78(3):427-35. doi: 10.1097/00000542-199303000-00005. PMID 8457043
- [Result] Benedetto M, Romano R, Baca G, Sarridou D, Fischer A, Simon A, Marczin N. Inhaled nitric oxide in cardiac surgery: Evidence or tradition? Nitric Oxide. 2015 Sep 15;49:67-79. doi: 10.1016/j.niox.2015.06.002. Epub 2015 Jul 14. PMID 26186889
- [Result] Clark RH, Kueser TJ, Walker MW, Southgate WM, Huckaby JL, Perez JA, Roy BJ, Keszler M, Kinsella JP. Low-dose nitric oxide therapy for persistent pulmonary hypertension of the newborn. Clinical Inhaled Nitric Oxide Research Group. N Engl J Med. 2000 Feb 17;342(7):469-74. doi: 10.1056/NEJM200002173420704. PMID 10675427
- [Result] Cornfield DN, Maynard RC, deRegnier RA, Guiang SF 3rd, Barbato JE, Milla CE. Randomized, controlled trial of low-dose inhaled nitric oxide in the treatment of term and near-term infants with respiratory failure and pulmonary hypertension. Pediatrics. 1999 Nov;104(5 Pt 1):1089-94. doi: 10.1542/peds.104.5.1089. PMID 10545552
- See also: Springer — http://link.springer.com/article/10.1007%2Fs00595-006-3226-5
- See also: biomed central — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3649943/
- See also: Nature Publishing Group — http://www.nature.com/nature/journal/v327/n6122/abs/327524a0.html
- See also: NEJM — http://www.nejm.org/doi/full/10.1056/NEJM200002173420704